CLINICAL TRIAL: NCT02428465
Title: Purposeful Parenting: Enhanced Anticipatory Guidance for the First Year of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Megan Bair-Merritt, Associate Professor of Pediatrics, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-33740
Record Dates: First submitted 2015-04-08; First posted 2015-04-28 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Parenting
Keywords: Purposeful Parenting; Parenting stress; Social-emotional and linguistic (SEL) skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purposeful Parenting (Experimental): Families randomized to the intervention group will receive their pediatric provider's usual anticipatory guidance plus Purposeful Parenting.
  Interventions: Behavioral: Purposeful Parenting
- Control Group (No Intervention): Families randomized to the control group will receive usual anticipatory guidance, delivered at the discretion of their pediatric provider, at each well-child visit in the first 12 months of life.

INTERVENTIONS:
Behavioral: Purposeful Parenting — Purposeful Parenting reinforces responsive interactions that help promote emerging developmental skills. This information is presented over the course of a child's first 12 months, such that core lessons are the same but specific skills are designed to be developmentally appropriate. This repetitiveness, along with the provision of age-appropriate behavioral guidance, will allow parents to successfully engage in responsive interactions with their children.
  Arms: Purposeful Parenting

SUMMARY:
Pediatricians' provision of parenting-focused anticipatory guidance often does not meet parents' needs; the few studies that have investigated primary-care based strategies to promote positive parenting rely on time-intensive, high-cost interventions, thereby limiting their generalizability. Therefore, the Purposeful Parenting was developed as a universal program of enhanced anticipatory guidance. At each well-child visit in the first year of a child's life, Purposeful Parenting provides parents with: 1) scripted anticipatory guidance and handouts focused on the child's emerging social-emotional and linguistic (SEL) skills, brain development and the importance of responsive parenting; and 2) a "reminder" item (e.g., a "Smile at Me" onesie) that allows for in-office role modeling and promotes practicing of an age-specific, nurturing parent-child interaction. If an in-office intervention is missed (e.g. parent cancels visit, interventionist out sick) the intervention will be delivered by telephone if possible by the site-based clinical interventionists and the "reminder" items will be mailed.

DETAILED DESCRIPTION:
The investigators will conduct a two-phase study. Phase I (months 1-4) will entail a brief pilot of Purposeful Parenting in three Boston-based health centers to optimize quality and logistical details. Phase II (months 5-36) will determine, with a parallel group randomized controlled trial (RCT), whether delivering Purposeful Parenting leads to increased responsive parenting at the intervention's conclusion (in intervention vs control parents), assessed using a validated observational measure. The investigators will enroll 260 low-income families with a full term newborn infant who present for well-child care. Families randomized to the control group will receive usual anticipatory guidance at each well-child visit in the first 12 months of life. Families randomized to the intervention group will receive usual anticipatory guidance plus Purposeful Parenting. As secondary outcomes, the investigators will explore the degree to which Purposeful Parenting (in intervention vs control parents) increases parental knowledge about responsive parenting and child development, reduces parenting stress and improves perceptions of parenting self-efficacy (via validated parental self-report measures) at the conclusion of the intervention. Investigators will explore potential differences by study group in child SEL development at the conclusion of the intervention. In addition, investigators will examine differences in the above listed outcomes are 6 months following the intervention. The RCT will include the collection of process level data including cost.

ELIGIBILITY:
Inclusion Criteria:

* Families (parent >=18 years of age) with a newborn, born at >= 34 weeks, presenting for well-child care
* Family plans to remain at that practice
* English or Spanish speaking

Exclusion Criteria:

* Debilitating chronic condition; prematurity (<34 weeks gestation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Responsive Parenting | At intervention conclusion (child is 12 months)
  Responsive parenting will be assessed using the Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLOTM), which involves an observer watching a 10 minute videotaped interaction to assess interaction between a parent and her infant or toddler. The PICCOLO is well-validated with inter-rater reliability=0.77; scale reliability=0.78; content, construct and predictive validity are acceptable.
Responsive Parenting | 6 months post intervention (child is 18 months)
  Responsive parenting will be assessed using the Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLOTM), which involves an observer watching a 10 minute videotaped interaction to assess interaction between a parent and her infant or toddler. The PICCOLO is well-validated with inter-rater reliability=0.77; scale reliability=0.78; content, construct and predictive validity are acceptable.

SECONDARY OUTCOMES:
Parental knowledge of infant/toddler development, health and safety, and positive parenting practices | At intervention conclusion (child is 12 months) and 6 months post intervention (child is 18 months)
  Parental knowledge of infant/toddler development, health and safety, and positive parenting practices will be assessed by the 75-item Knowledge of Infant Development (KIDI) scale. The scale was developed to be accessible to parents with limited literacy and to be culturally neutral. Cronbach's alpha for parents is 0.82; test-retest reliability for parents is 0.92; validity has also been deemed acceptable.
Parenting stress | At intervention conclusion (child is 12 months) and 6 months post intervention (child is 18 months)
  Parenting stress will be assessed by the 36-item short form of the Abidin's Parenting Stress Index (PSI), with subscales including perceptions of social isolation, attachment to the child and parental health. Cronbach's alpha is 0.91 for the total scale; six month test-retest coefficients are 0.68-0.85.
Satisfaction and confidence in parenting skills | At intervention conclusion (child is 12 months) and 6 months post intervention (child is 18 months)
  Satisfaction and confidence in parenting skills will be assessed by the 17-item Parenting Sense of Competency scale. Internal reliability is excellent, with Cronbach's alphas ranging from 0.75-0.88. Two sub-scales measure perceptions of efficacy and satisfaction in the parenting role.

OTHER OUTCOMES:
Social and emotional competence | At intervention conclusion (child is 12 months) and 6 months post intervention (child is 18 months)
  Social and emotional competence will be assessed by the 42-item Brief Infant-Toddler Social and Emotional Assessment (BITSEA). Cronbach's alpha is 0.76, and test-retest reliability is 0.61-0.75. The measure correlates well with the Child Behavior Checklist.
Child language and communication skills | At intervention conclusion (child is 12 months) and 6 months post intervention (child is 18 months)
  Parent report of child language and communication skills will be assessed by the MacArthur-Bates Communicative Development Inventories (CDI). The CDI: Words and Gestures, used for children between the ages of 8 and 18 months, documents the child's understanding of early vocabulary items both understood and used, and records the communicative and symbolic gestures. The CDI: Words and Sentences, used for children between the ages of 16 and 30 months, documents the child's production and use of words and analyzes the early phases of grammar. The CDI has excellent test-retest reliability, concurrent validity and correlates well with other measures of child language development.
Cost | Collected for duration of the intervention (12 months of intervention per child)
  Cost data (e.g., staff time and training; supplies and materials) collected to assess marginal cost of intervention
Barriers and Facilitators to Intervention Sustainability | Interviews conducted once at 36 months (study conclusion)
  Qualitative interviews with key stakeholders about barriers and facilitators of sustaining intervention

CONTACTS AND LOCATIONS:
Overall Officials: Megan H Bair-Merritt, MD, MSCE, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Dimock Health Center, Roxbury, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coker TR, Windon A, Moreno C, Schuster MA, Chung PJ. Well-child care clinical practice redesign for young children: a systematic review of strategies and tools. Pediatrics. 2013 Mar;131 Suppl 1(Suppl 1):S5-25. doi: 10.1542/peds.2012-1427c. PMID 23457149
- [Background] Magar NA, Dabova-Missova S, Gjerdingen DK. Effectiveness of targeted anticipatory guidance during well-child visits: a pilot trial. J Am Board Fam Med. 2006 Sep-Oct;19(5):450-8. doi: 10.3122/jabfm.19.5.450. PMID 16951294
- [Background] Olson LM, Inkelas M, Halfon N, Schuster MA, O'Connor KG, Mistry R. Overview of the content of health supervision for young children: reports from parents and pediatricians. Pediatrics. 2004 Jun;113(6 Suppl):1907-16. PMID 15173461
- [Background] Cook GA, Innocenti MS, Roggman LA, Jump Norman VK. PICCOLO: A simple parent-child interaction measure and its use in early intervention. New York, 2011.
- [Background] Kruizinga I, Jansen W, Mieloo CL, Carter AS, Raat H. Screening accuracy and clinical application of the Brief Infant-Toddler Social and Emotional Assessment (BITSEA). PLoS One. 2013 Aug 30;8(8):e72602. doi: 10.1371/journal.pone.0072602. eCollection 2013. PMID 24023626
- [Background] Rescorla L, Alley A. Validation of the language development survey (LDS): a parent report tool for identifying language delay in toddlers. J Speech Lang Hear Res. 2001 Apr;44(2):434-45. doi: 10.1044/1092-4388(2001/035). PMID 11324663
- [Background] MacPhee D. Knowledge of infant development inventory. Chapel Hill, NC: University of North Carolina; 1981.
- [Background] Abidin R. Parenting Stress Index: Professional Manual. 3rd ed. Odessa, FL: Psychological Assessment Resources; 1995.
- [Background] Gilmore L, Cuskelly M. Factor structure of the Parenting Sense of Competence scale using a normative sample. Child Care Health Dev. 2009 Jan;35(1):48-55. doi: 10.1111/j.1365-2214.2008.00867.x. Epub 2008 Oct 22. PMID 18991983